CLINICAL TRIAL: NCT02803749
Title: The Tolerability of Buspirone for the Treatment of Anxiety in Parkinson's Disease
Brief Title: Buspirone in Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Irene Richard, Professor of Neurology, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 61141
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Parkinson Disease; Anxiety
MeSH Terms: conditions — Parkinson Disease; Anxiety Disorders | interventions — Buspirone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buspirone (Experimental): Flexible dosage buspirone (maximum dosage 30 mg twice daily) for 12 weeks.
  Interventions: Drug: Buspirone
- Placebo (Placebo Comparator): Flexible dosage placebo for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buspirone
  Arms: Buspirone
Drug: Placebo
  Arms: Placebo

SUMMARY:
Anxiety is highly prevalent in Parkinson's disease and negatively impacts quality of life yet it frequently remains untreated and there have been no clinical trials dedicated to evaluating the pharmacological treatment of anxiety in Parkinson's disease. Buspirone is effective for the treatment of generalized anxiety disorder in the general and elderly population. It is not known if it is effective for the treatment of anxiety in Parkinson's disease. This is a single-center, placebo-controlled, double-blind design with participants randomized with a 4:1 allocation ratio to flexible dosage buspirone (maximum dosage 30 mg twice daily) or placebo for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD by UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria
* Significant anxiety as determined by the self-rated Parkinson Anxiety Scale (score ≥ 14)
* Able to provide written informed consent
* At least 18 years of age

Exclusion Criteria:

* Diagnosis of atypical or secondary parkinsonism
* Concomitant treatment with an MAO inhibitor within the 14 days prior to screening visit
* Significant renal or hepatic impairment
* Significant cognitive impairment defined as MOCA score < 23
* On-going depression with suicidal or homicidal ideation and concern for patient safety based on clinical determination by the investigator
* Allergy or intolerance to study drug, matching placebo, or their formulations
* History of prior exposure to study drug
* Lactating or pregnant woman
* Concomitant treatment with a disallowed medication (detailed in section 6.2)
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
* Concomitant treatment with an anxiolytic or antidepressant will be allowed however potential participants who had dosage changes in the 30 days prior to the screening visit will be excluded
* Use of an investigational drug within 30 days prior to screening visit
* Any medical or psychiatric comorbidity that, in the opinion of the investigator, would compromise study participation
* Dysphagia defined as a score of ≥ 2 on MDS-UPDRS Item 2.3 Chewing and Swallowing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-10; Primary Completion 2019-01 (Actual); Study Completion 2019-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Richard, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Buspirone: Flexible dosage buspirone (maximum dosage 30 mg twice daily) for 12 weeks.
  Buspirone
- Placebo: Flexible dosage placebo for 12 weeks.
  Placebo
Period: Overall Study
Arm/Group | Buspirone | Placebo
Started | 17 | 4
Completed | 12 | 4
Not Completed | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buspirone | Placebo | Total
Number analyzed (Participants) | 17 | 4 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (9.8) | 70.3 (10.6) | 66.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 13 | 1 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 16 | 4 | 20
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 4 | 21
Married participants [Count of Participants; unit: Participants] | 14 | 4 | 18
Greater than high school education [Count of Participants; unit: Participants] | 14 | 4 | 18
History of Depression [Count of Participants; unit: Participants] | 2 | 1 | 3
Taking Antidepressant or Anxiolytic [Count of Participants; unit: Participants] | 15 | 2 | 17
Hoehn and Yahr Stage [Count of Participants; unit: Participants] — The Hoehn and Yahr scale defines broad categories of motor function in Parkinson's disease with a score of 1 indicating Unilateral involvement, a score of 2 indicating Bilateral involvement without balance impairment, a score of 3 indicating mild-moderate disability with balance impairment and a score of 4 indicating severe disability, still able to walk or stand unassisted.
  Participants
    1 | 3 | 0 | 3
    2 | 11 | 3 | 14
    3 | 3 | 0 | 3
    4 | 0 | 1 | 1
MDS-UPDRS [Mean (Standard Deviation); unit: units on a scale] — The Movement Disorder Society Unified Parkinson's Disease Rating scale evaluates aspects of motor and non-motor experiences of daily living. The scale assesses non-motor experiences of daily living (NM-EDL; range 0-52), motor experiences of daily living (M-EDL; range 0-52), motor examination ; range 0-132), and motor complications (range 0-24). Each subscale has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. Scores for sub scales are summed to create the Total score. The total range of scores is 0-260. Higher scores mean worse outcomes.
  units on a scale
    Total | 59.6 (22.5) | 67.5 (24.3) | 61.1 (22.4)
    nM-EDL | 11.4 (5.2) | 13 (5.2) | 11.7 (5.1)
    M-EDL | 12.9 (7.6) | 14.5 (7.5) | 13.2 (7.4)
    Motor | 32.3 (15.3) | 37.5 (11.7) | 33.3 (14.5)
    Motor Compications | 3.0 (3.3) | 3.3 (3.5) | 3.1 (3.2)
Unified Dyskinesia Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The Unified Dyskinesia Rating Scale captures the essential features of dyskinesia in Parkinson's disease within a single scale, including patient perceptions, time factors, anatomical distribution, objective impairment, severity, and disability. A lower score is a better outcome for this measure.
  units on a scale | 5.2 (7.3) | 3.8 (5.2) | 5.0 (6.9)
Parkinson Anxiety Scale [Mean (Standard Deviation); unit: units on a scale] — The Parkinson's Anxiety Scale measures the anxiety of Participants on a scale of 0-48 with a lower score being a better outcome.
  units on a scale | 19.1 (3.9) | 19.3 (5.1) | 19.1 (4.0)
Hamilton Anxiety Scale [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Anxiety Scale is used to measure the severity of anxiety symptoms. The scale ranges from 0-56 with a lower score being the desired outcome.
  units on a scale | 11.4 (4) | 12.3 (2.9) | 11.5 (3.7)
Hospital Anxiety and Depression Scale - Anxiety [Mean (Standard Deviation); unit: units on a scale] — The Hospital Anxiety and Depression Scale is a fourteen item scale consisting of seven depression and seven anxiety questions. The scores range from 0-42 (for 14 questions) and 0-21 for each subsection of anxiety and depression. For the purposes of this information, anxiety and depression scores are split up with this data showing anxiety results so the scale ranges from 0-21 with a low score being better.
  units on a scale | 8.2 (3.1) | 6.8 (3.1) | 7.9 (3.0)
Hospital Anxiety and Depression Scale - Depression [Mean (Standard Deviation); unit: units on a scale] — The Hospital Anxiety and Depression Scale is a fourteen item scale consisting of seven depression and seven anxiety questions. The scores range from 0-42 (for 14 questions) and 0-21 for each subsection of anxiety and depression For the purposes of this information, anxiety and depression scores are split up with this data showing depression results so the scale ranges from 0-21 with a low score being better.
  units on a scale | 5.4 (3.1) | 4.8 (2.6) | 5.2 (3.0)
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA) measures cognitive capacity on a scale of 0-30 with a higher score being the better outcome.
  units on a scale | 26.3 (2.3) | 26.8 (2.1) | 26.4 (2.2)
Started Taking Antidepressant or Anxiolytic during Study [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Fail to Complete the 12-week Study on Study Drug.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 17 | 4
Participants | 7 | 0

2. Secondary Outcome: Mean Change in Hamilton Anxiety Rating Scale (HAM-A) From Baseline to 12 Weeks
Description: The HAM-A assess anxiety on 0-56 scale where a higher score represents a higher level of anxiety.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 12 | 4
score on a scale | -4.21 (1.13) | -3.36 (1.97)

3. Secondary Outcome: Number of Responders (>50% Reduction From Baseline or Reduction to ≤7 on HAM-A) at 12 Weeks
Description: The HAM-A assess anxiety on 0-56 scale where a higher score represents a higher level of anxiety.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 12 | 4
Participants | 9 | 1

4. Secondary Outcome: Number of "Much Improved" or "Very Much Improved" on Patient Global Impressions-Improvement (PGI-I) at 12 Weeks
Description: The PGI-I assesses patient global impression of improvement on a 7-point scale where 1 = "very much improved" and 7 = "very much worse."
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 12 | 4
Participants | 3 | 0

5. Secondary Outcome: Mean Change in Anxiety Using the Hospital Anxiety and Depression Scale (HADS)
Description: The HADS assesses anxiety on a scale of 0-21 and depression on a scale of 0-21 with higher scores indicating higher levels of anxiety and depression respectively.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 12 | 4
score on a scale | -1.87 (0.98) | -0.89 (1.71)

6. Secondary Outcome: Mean Change in Unified Dyskinesia Rating Scale (UDysRS) From Baseline to 12 Weeks
Description: The UDysRS assesses dyskinesias on a scale of 0-104 where a higher score represents more severe dyskinesias.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 12 | 4
score on a scale | .72 (3.22) | 7.78 (6.44)

7. Secondary Outcome: Number of "Much Improved" or "Very Much Improved" on Clinical Global Impressions-Improvement (CGI-I) at 12 Weeks
Description: The CGI-I assesses clinician global impression of improvement on a 7-point scale where 1 = "very much improved" and 7 = "very much worse."
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 12 | 4
Participants | 5 | 2

8. Secondary Outcome: Mean Change in Hospital Anxiety and Depression Scale (HADS) - Depression From Baseline to 12 Weeks
Description: as for outcome 5
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 12 | 4
units on a scale | -.95 (.46) | .34 (.81)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Buspirone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/4
Other Adverse Events (participants affected / at risk) | 5/17 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Buspirone (N=17) | Placebo (N=4)
Increased freezing of gait (General disorders) | 5 | 0
tremor (General disorders) | 3 | 0
sleep difficulties (General disorders) | 2 | 2
dizziness (General disorders) | 2 | 0
increased fatigue (General disorders) | 2 | 0
increased tremor (General disorders) | 1 | 3
balance impairment (General disorders) | 1 | 2
increased peripheral edema (General disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Gait Difficulties (General disorders) | 0 | 1
Vertigo (General disorders) | 0 | 1
Vision Changes (Eye disorders) | 0 | 1
Weakness (General disorders) | 0 | 1
Bradycardia (General disorders) | 1 | 0
Constipation (General disorders) | 1 | 0
Dysphagia (General disorders) | 1 | 0
Fuzziness (General disorders) | 1 | 0
Gastritis/Duodenitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Illness (Gastrointestinal disorders) | 1 | 0
Hand Cramps (General disorders) | 1 | 0
Headache (General disorders) | 1 | 0
Increased agitation (General disorders) | 1 | 0
Increased appetite (General disorders) | 1 | 0
Increased balance impairment (General disorders) | 1 | 0
Increased dystonia (General disorders) | 1 | 0
Increased irritability (General disorders) | 1 | 0
Increased Knee pain (General disorders) | 1 | 0
Increased OFF time (General disorders) | 1 | 0
increased pain secondary to lipomas (General disorders) | 1 | 0
insomnia (General disorders) | 1 | 0
joint stiffness (General disorders) | 1 | 0
Left shoulder/neck pain (General disorders) | 1 | 0
leg pain (General disorders) | 1 | 0
nasal congestion (General disorders) | 1 | 0
numbness (General disorders) | 1 | 0
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-05-27): https://cdn.clinicaltrials.gov/large-docs/49/NCT02803749/Prot_SAP_000.pdf
  • Informed Consent Form (2016-06-09): https://cdn.clinicaltrials.gov/large-docs/49/NCT02803749/ICF_001.pdf